CLINICAL TRIAL: NCT05695313
Title: Phase II Multicentric, Randomized Study Versus Placebo for the Prevention of Neurotoxicity Induced by Weekly PACLITAXEL
Brief Title: Randomized Study Versus Placebo for the Prevention of Neurotoxicity Induced by Weekly PACLITAXEL
Acronym: NEUROTAX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-A01940-43
Record Dates: First submitted 2023-01-02; First posted 2023-01-25 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: breast; neuropathy; OnLife; dietary supplement; Paclitaxel
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Standard chemotherapy PACLITAXEL + placebo dietary supplement
  Interventions: Other: Placebo
- OnLife® (Experimental): Standard chemotherapy + OnLife® dietary supplement
  Interventions: Drug: OnLife®

INTERVENTIONS:
Drug: OnLife® — It is administered for the duration of PACLITAXEL chemotherapy with the first administration performed 5 days before the first PACLITAXEL administration. The OnLife supplement will be continued for another 4 weeks after the last PACLITAXEL administration.
  One tablet in the morning and one in the evening daily
  Arms: OnLife®
Other: Placebo — It is administered for the duration of PACLITAXEL chemotherapy with the first administration performed 5 days before the first PACLITAXEL administration. Placebo will be continued for another 4 weeks after the last PACLITAXEL administration.
  One tablet in the morning and one in the evening daily
  Arms: Placebo

SUMMARY:
This study recommends the use of OnLife dietary supplement, which will be followed by a few day before the initiation of PACLITAXEL, for the prevention of PACLITAXEL induced neuropathy. OnLife will be continued one month after stopping chemotherapy.

This would limit the number of PACLITAXEL dose reductions and premature interruptions of this chemotherapy, thus potentially improving the results in terms of antitumor efficacy, while improving the quality of life of patients treated with weekly PACLITAXEL.

DETAILED DESCRIPTION:
This study recommends the use of OnLife dietary supplement which will be followed by a few day before the initiation of PACLITAXEL for the prevention of PACLITAXEL induced neuropathy. OnLife will be continued one month after stopping chemotherapy. This would limit the number of PACLITAXEL dose reductions and premature interruptions of this cehemotherapy, thus potentially improving the results in terms of antitumor efficacy while improving the quality of life of patients treated with weekly PACLITAXEL.

Two treatment arms :

- ARM A : 20 patients included in the placebo arm (Standard chemotherapy with PACLITAXEL + placebo dietary supplement) ARM B : 40 patients included in the experimental arm (standard PACLITAXEL chemotherapy + OnLife® food supplement)

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patient with neo-adjuvant or adjuvant management, with an indication for weekly PACLITAXEL 80 mg/m² for 12 courses.
* Age ≥ 18 years
* Performans Status ≤ 3 according to Karnofsky and life expectancy greater than 6 months
* For patients of childbearing age, effective contraception while taking Onlife®/placebo.
* Patient able to swallow OnLife/placebo® tablets easily
* Patient able and willing to follow all study procedures (including the completion of numerous questionnaires) in accordance with the protocol
* Patient has understood, signed and dated the consent form
* Patient affiliated to the social security system

Exclusion Criteria:

* Patient previously started on PACLITAXEL
* Known allergy to any of the substances in the study product Onlife®/placebo (fish oil product)
* Diabetes
* Exogenous (Alcoholism)
* History of peripheral neuropathy at inclusion and/or presence of sensory and/or motor disorders due to other neurological diseases
* Pregnant or breastfeeding woman
* Other uncontrolled progressive pathologies
* Impossible or random follow-up
* Persons deprived of liberty or under guardianship (including curatorship)
* Inability to submit to the medical follow-up of the trial for geographical, social or psychological reasons.

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Neuropathies will be graded by the oncologist using the NCI-CTCAE version 5.0. | At 3 months
  Neuropathies will be graded by the oncologist using the NCI-CTCAE version 5.0. during the consultation with the oncologist at 3 months.
  The AE graded from 1 to 5. Grade 1 is a better and grade 5 is a worst outcome.

SECONDARY OUTCOMES:
Evaluation of Neuropathic pain symptom inventory (NPSI) scores | At 12 weeks, 16 weeks, 6 months and 12 months
  Evaluation of Neuropathic pain symptom inventory scores by the questionnaire. The minimum value is 0 (no pain) and the maximum value is 10 (maximum pain)
All peripheral neuropathies graded by the oncologist according to CTCAE V5.0 | Every 4 weeks for one year
  Assess the rate of grade ≥ 2 peripheral neuropathy by NCI-CTCAE V5.0 The AE graded from 2 to 5. Grade 2 is a better and grade 5 is a worst outcome.
Time to onset of grade ≥ 2 neuropathy. | During 1 year
  Assess time to onset of grade ≥ 2 neuropathy by Kaplan-Meyer method The AE graded from 2 to 5. Grade 2 is a better and grade 5 is a worst outcome.
Number of toxicities attributable to OnLife® dietary supplement | Every 4 weeks for one year
  Assess toxicities attributable to OnLife® dietary supplement by NCI-CTCAE V5.0
Number of participants with musculoskeletal and joint pain | At 12 weeks, 16 weeks 6 months and 12 months.
  Musculoskeletal and joint pain will be defined and graded according to the CTCAE v5.0 classification
Compliance with the Onlife®/Placebo dietary supplement | 16 weeks
  Compliance with the Onlife®/Placebo dietary supplement will be assessed by the accounting for treatments returned by patients to the pharmacy.
Quality of life of participants | At baseline and then every 4 weeks for 4 months and then at 6 and 12 months.
  Quality of life will be assessed by the EORTC QLQ C30 self-questionnaires and its associated module Chemotherapy-Induced Peripheral Neuropathy (CIPN 20).
  The minimum value is 1 (no way) and the maximum value is 4 (a lot)
The number and rate of women with at least one dose reduction due to peripheral neuropathy. | During 1 year
  By NCI-CTCAE V5.0
Name of all concomitant treatments administered for neuropathy | At 12 weeks, 16 weeks, 6 months and 12 months.
  By recording data in the eCRF for both arms
Evaluation of Overall Neuropathy Limitations Scale (ONLS) scores | At 12 weeks, 16 weeks, 6 months and 12 months
  Evaluation of ONLS scores by the questionnaires. The minimum value is 0 (better outcome) and the maximum value is 5 (worse outcome)
Compliance with the Onlife®/Placebo dietary supplement | 16 weeks
  Compliance with the Onlife®/Placebo dietary supplement will be assessed by the Morisky questionnaire
The number and rate of women with at least one discontinuation of PACLITAXEL due to peripheral neuropathy. | During 1 year
  By NCI-CTCAE V5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc, Dijon, France